CLINICAL TRIAL: NCT07294248
Title: Diagnostic Role of Magnetic Resonance Imaging and Ultrasonography in Characterization of Superficial Soft Tissue Masses.
Brief Title: Role of MRI and US in Superficial Soft Tissue Masses
Acronym: MRI/US in SSTM
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Sobhy Aziz, Resident, Sohag University
Other Study IDs: Soh-Med--25-11-15MS
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Superficial Soft Tissue Masses
MeSH Terms: interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with superficial soft tissue masses: Participants diagnosed with superficial soft tissue masses undergoing ultrasound and MRI for diagnostic characterization.
  Interventions: Other: Diagnostic imaging (US and MRI).

INTERVENTIONS:
Other: Diagnostic imaging (US and MRI). — Ultrasonography and MRI are performed as part of routine diagnostic evaluation, these are not therapeutic interventions

SUMMARY:
The goal of this observational study to evaluate the accuracy of Magnetic Resonance Imaging and Ultrasonography in characterization of superficial soft tissue masses.

DETAILED DESCRIPTION:
This study is a prospective observational study aiming to evaluate and compare the diagnostic roles of magnetic resonance imaging (MRI) and ultrasound (US) in the characterization of superficial soft tissue masses. The study will be conducted in [ Sohag ] over a period of [ 6 Months].

Participants Consecutive patients presenting with superficial soft tissue masses (located within the subcutaneous tissue. Inclusion criteria include Patients who suffer from superficial soft tissue lesions measurable by both MRI and US in both sex and of any age group, will be included in the study , Exclusion criteria include Patients unwilling to complete study, Patients with absolute or relative contraindications for imaging including; claustrophobia, metallic implants, pacemaker and prosthetic heart valves for MRI, will be evaluated by US.

Objectives

* Primary objective: To determine the added value of MRI compared with ultrasound in accurate characterization of superficial soft tissue masses (benign vs malignant features).
* Secondary objectives:
* Assess concordance between MRI and US in differentiating cystic versus solid lesions.
* Identify specific imaging features on MRI and US that best predict malignant potential.
* Evaluate interobserver agreement for MRI and US interpretations.

Methods Imaging Protocols

* Ultrasound: High-resolution ultrasound with Doppler will be performed to assess size, echotexture, margins, internal septations, vascularity, and presence of calcifications. Lesions will be categorized as solid, cystic, or complex.
* MRI: MRI protocols will include T1-weighted, T2-weighted, STIR, and post-contrast sequences, with assessment of lesion margins, internal composition, enhancement pattern, diffusion characteristics where available, and involvement of adjacent structures.

Data Collection and Outcomes

* Demographic data, lesion characteristics (size, location, depth), imaging features, and final diagnosis will be recorded.
* Primary outcome: Diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) of MRI and US individually and in combination for distinguishing malignant from benign masses.
* Secondary outcomes: Agreement between modalities; correlation of specific imaging features with histopathology if available.

Data Analysis The collected data will be statistically analyzed using SPSS. Chi-square (X2 analysis) contingency analysis will be used. Results will be discussed. Conclusions and recommendations will be suggested based on the results.

Ethical Considerations

- The study will be conducted in accordance with the Declaration of Helsinki. Informed consent will be obtained from all participants. The study protocol has been or will be approved by the [Institutional Review Board/Ethics Committee].

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from superficial soft tissue lesions in both sex and of any age group, will be included in the study.

Exclusion Criteria:

* Patients unwilling to complete study.
* Patients with absolute or relative contraindications for imaging including; claustrophobia, metallic implants, pacemaker and prosthetic heart valves for MRI, will be evaluated by US.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with clinically or radiologically suspected superficial soft tissue masses who are referred for diagnostic ultrasound and MRI evaluation at the hospital during the study period. The study population includes adults and children meeting the eligibility criteria and undergoing imaging as part of routine diagnostic assessment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Ultrasound and MRI in characterization of superficial soft tissue masses. | During initial diagnostic assessment
  Evaluation of the ability of ultrasound and MRI to correctly characterize superficial soft tissue masses. Diagnostic accuracy measures will include sensitivity, specificity, positive predictive value, and negative predictive value compared to the final reference diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hassan Alam-Eldeen, MD, Principal Investigator
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy and confidentiality considerations